CLINICAL TRIAL: NCT02485951
Title: Big-bubble Deep Anterior Lamellar Keratoplasty: Central Versus Peripheral Air Injection
Brief Title: Central Versus Peripheral Air Injection for DALK (Deep Anterior Lamellar Keratoplasty)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sepehr Feizi, MD, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShaheedBMU54
Record Dates: First submitted 2015-06-13; First posted 2015-06-30 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2015-06

CONDITIONS: Keratoconus
Keywords: deep anterior lamellar keratoplasty; big-bubble technique; peripheral air injection; keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Central air injection (Active Comparator): The needle was moved radially inside the trephination site and advanced to the central or paracentral cornea.
  Interventions: Procedure: Central air injection
- Peripheral air injection (Active Comparator): The needle was inserted into the deep stroma from the trephination site and advanced into the peripheral cornea to approximately 1.5 mm anterior to the limbus.
  Interventions: Procedure: Peripheral air injection

INTERVENTIONS:
Procedure: Central air injection — Air was injected inside the trephination site in the central injection group.
  Arms: Central air injection
Procedure: Peripheral air injection — Air was injected at the corneal periphery outside the trephination site.
  Arms: Peripheral air injection

SUMMARY:
Different techniques of deep anterior lamellar keratoplasty (DALK) have been introduced to create a uniform recipient bed, thereby reducing complications, such as interface irregularity and opacification encountered with conventional lamellar keratoplasty. The big-bubble technique provides a planned, safe, quick and consistent baring of Descemet membrane (DM) by injection of air deep into the stroma. Nevertheless, this technique has a long learning curve with a low success rate of big-bubble formation and a high rate of DM perforation when performed by surgeons in training. Different modifications to the original technique using intraoperative instruments such as corneal pachymetry, anterior segment optical coherence tomography (OCT), and femtosecond laser, have been used to increase the chances of achieving a successful DM detachment from the deep stroma by air injection. Even with these innovations, the rate of successful big-bubble formation did not reach 100%. Recently, the investigators described a modification to the original big-bubble DALK in which a 27-gauge needle was inserted into the stroma peripherally from the trephination site towards the limbus. The investigators found that air injection peripheral to the trephination can effectively and reproducibly separate the corneal stroma from the Descemet membrane (DM). This study was aimed to compare the success rate and complications of big-bubble DALK using central versus peripheral air injection performed by senior cornea fellows under the supervision of an experienced faculty member in an academic hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate (48 D < mean keratometry < 55 D) to advanced (mean keratometry ≥ 55 D or immeasurable keratometry) keratoconus were enrolled.

Exclusion Criteria:

* History of ocular surgery, concomitant ocular pathologies, such as vernal keratoconjunctivitis, cataract, glaucoma, and retinal abnormalities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The rate of successful big-bubble formation | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran